CLINICAL TRIAL: NCT03704285
Title: Development of Pharmacokinetic / Pharmacodynamic (pk/pd) Model of Propofol in Patients With Severe Burns
Brief Title: Development of pk/pd Model of Propofol in Patients With Severe Burns
Acronym: HUAPQ
Status: Terminated | Type: Observational
Why Stopped: Outbreak COVID 19
Sponsor: Victor Contreras, MSN (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor-Investigator, Victor Contreras, MSN, Co-Investigator. Project Manager of Department of Anesthesiology, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Other Study IDs: 171215006
Record Dates: First submitted 2018-10-03; First posted 2018-10-12 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia; Burned; Operative Wound
Keywords: anesthesia; burned; TIVA; propofol
MeSH Terms: conditions — Burns; Surgical Wound | interventions — Propofol; Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Propofol: Severe burn adult under general anesthesia with propofol + remifentanil evaluation of propofol effect using BIS
  Interventions: Drug: Propofol; Device: BIS

INTERVENTIONS:
Drug: Propofol — Patients undergoing general anesthesia using target controlled infusion of propofol. Initial bolus of 1-2 mg/kg and then a continuous infusion of 10 mg/kg/hr that will be adjusted adjusted to maintain a BIS between 40 and 60.
  Other Names: Propofol Intravenous dose
Device: BIS — GeneralAnesthesia maintenance with propofol+remifentanil guided by BIS monitoring.
  Other Names: General anesthetic

SUMMARY:
Burn injuries are a prevalent problem. Actually, in Chile the Ministry of Health has recorded 6435 hospital burns and has reported 569 deaths from this cause. The specific mortality rate for burning in Chile was 4.5 per 100,000 inhabitants per year. Survival in extensive burns has progressively improved, thanks to advances in understanding the pathophysiology of the burn and its more aggressive treatment. This requires effective prehospital treatment, transportation, resuscitation, support of vital functions and repair of the skin cover.

Much of the procedures performed in large burns require general anesthesia. Being Total Intravenous Anesthesia (TIVA) with propofol an alternative that would have advantages over inhalational anesthesia, as a decrease in postoperative nausea and vomiting and produce less environmental pollution 3 and the antihyperalgesic effect of propofol. Within TIVA - Target Control Infusion (TCI) - uses infusion systems that incorporate PK-PD models for predict the dose of drug required to reach a certain concentration in the target organ.

The formulation of a PK model that considers the variables of this group of patients, such as: degree of injury, inflammatory state and compromised body surface; associated with general variables such as: age, weight and nutrition, it would allow to reduce the predictive error in this population, thus improving the dosing of these patients when using TCI.

Given the lack evidence on the PK-PD of propofol is this group of patients burned, has led to raise the development of this study that seeks to develop a PK-PD model that fits them.

DETAILED DESCRIPTION:
Patients will be invited to participate before surgery, the inclusion criteria will be revised and the informed consent will be signed.

In the operating room will be recorded demographic data and relevant background such as: Age, Weight, Size, BMI, Lean Mass, Fat Mass and Total body water among others.

Afterwards, in the operating room, the patient will be monitored regularly: ECG (DII) if feasible and pulse oximetry. An arterial catheter will be installed for monitoring and taking blood samples during the intraoperative period.

In addition, the EEG will be monitored through a frontal electroencephalographic monitoring (BIS) system; that will be recorded throughout the surgery.

The anesthetic induction will be with propofol and remifentanil. The propofol will be administered using an initial bolus of 1-2 mg / kg according to the criteria of the anesthetist and then a continuous infusion of 10 mg / kg / hr that will be adjusted adjusted to maintain a BIS between 40 and 60.

Plasma samples of propofol: arterial samples of 3-4 ml will be taken at 2, 5, 10, 30, 60 and/or 120 min after beginning the administration of propofol. Subsequently samples will be taken at 0, 5, 15, 30, 60, 120, 240 min and at 6-12 hrs after stopping the infusion of propofol. The samples will be centrifuged and stored at -20 ° C until analysis by HPLC.

ELIGIBILITY:
Inclusion Criteria:

* Severe burns with life risk that require treatment in Burn Units and / or Critical Patient Units.
* In spontaneous ventilation
* SAS 4

Exclusion Criteria:

* Electric burns
* ASA IV o V
* Inability to install BIS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Major burns
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Propofol plasmatic levels Measured by high pressure liquid chromatography | From start of propofol infusion to 12 hrs after stopped infusion of propofol.
  Propofol total dose. 2, 5, 10, 30, 60 and 120 min after induction with propofol. Subsequently, samples will be taken at 0, 5, 15, 30, 60, 120, 240 min and at 6-12 hrs after stopping infusion of propofol.

SECONDARY OUTCOMES:
Hemodynamics | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Arterial pressure (mmHg)
Heart Rate | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Heart rate (bpm)
Pulse oximetry | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  % oximetry saturation
BIS | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Depth of anesthesia will be recorded with BIS monitor. From 60 - 40

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortinez, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Victor Contreras, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Shin SW, Cho AR, Lee HJ, Kim HJ, Byeon GJ, Yoon JW, Kim KH, Kwon JY. Maintenance anaesthetics during remifentanil-based anaesthesia might affect postoperative pain control after breast cancer surgery. Br J Anaesth. 2010 Nov;105(5):661-7. doi: 10.1093/bja/aeq257. Epub 2010 Sep 28. PMID 20876698
- [Background] Cortinez LI, De la Fuente N, Eleveld DJ, Oliveros A, Crovari F, Sepulveda P, Ibacache M, Solari S. Performance of propofol target-controlled infusion models in the obese: pharmacokinetic and pharmacodynamic analysis. Anesth Analg. 2014 Aug;119(2):302-310. doi: 10.1213/ANE.0000000000000317. PMID 24977639
- [Background] Cortinez LI, Anderson BJ, Penna A, Olivares L, Munoz HR, Holford NH, Struys MM, Sepulveda P. Influence of obesity on propofol pharmacokinetics: derivation of a pharmacokinetic model. Br J Anaesth. 2010 Oct;105(4):448-56. doi: 10.1093/bja/aeq195. Epub 2010 Aug 14. PMID 20710020
- [Background] Eleveld DJ, Colin P, Absalom AR, Struys MMRF. Pharmacokinetic-pharmacodynamic model for propofol for broad application in anaesthesia and sedation. Br J Anaesth. 2018 May;120(5):942-959. doi: 10.1016/j.bja.2018.01.018. Epub 2018 Mar 12. PMID 29661412
- [Background] Rolle A, Paredes S, Cortinez LI, Anderson BJ, Quezada N, Solari S, Allende F, Torres J, Cabrera D, Contreras V, Carmona J, Ramirez C, Oliveros AM, Ibacache M. Dexmedetomidine metabolic clearance is not affected by fat mass in obese patients. Br J Anaesth. 2018 May;120(5):969-977. doi: 10.1016/j.bja.2018.01.040. Epub 2018 Mar 28. PMID 29661414